CLINICAL TRIAL: NCT07013968
Title: Healing Within: Smoking Cessation Intervention for American Indian Women Experiencing Intimate Partner Violence
Brief Title: Healing Within: Mindfulness Smoking Cessation Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Jeffrey A Henderson, MD, MPH, PI/Program Director, Black Hills Center for American Indian Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1 S06 GM146079-01-RP1; 1S06GM146079-01 (NIH)
Record Dates: First submitted 2023-05-10; First posted 2025-06-10 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Smoking Cessation
Keywords: Trauma-informed; Culturally tailored
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 48 Northern Plains Tribal women smokers who have experienced Intimate Partner Violence (IPV). (Experimental): These participants will experience a culturally tailored, trauma-informed mindfulness smoking cessation intervention.
  Interventions: Behavioral: culturally tailored, trauma-informed mindfulness smoking cessation intervention

INTERVENTIONS:
Behavioral: culturally tailored, trauma-informed mindfulness smoking cessation intervention — Eight weekly in-person group sessions, each 90 minutes long. From the second half of PY01 to PY04, sessions will be performed in closed in groups of 7-10 participants (with a total of 6 groups). The curriculum is grounded in Lakota values and trauma-informed care. Each of the eight sessions will begin and end with a Lakota serenity prayer and "wazílya" (smudging of sage), and the meaning and relevance of one of the Lakota values will be discussed. Through a storytelling approach, which is central to Lakota culture, the participants will learn about their value as a Lakota woman, the role of caŋṡaṡa, the association between unresolved trauma and smoking, and the importance of Lakota mind-based and mindfulness strategies in their lives.

SUMMARY:
Using a highly participatory approach, this study will assess the feasibility, acceptability, and satisfaction with a culturally tailored, trauma-informed smoking cessation intervention for Northern Plains Tribal women who have experienced intimate partner violence. If successful, other American Indian Tribes and Tribal communities can adapt this innovative smoking cessation curriculum for their communities.

DETAILED DESCRIPTION:
Cigarette smoking and intimate partner violence (IPV) are preventable, major public health concerns that result in severe physical and psychological consequences. Women who have experienced IPV are more likely to suffer from substance use, depression, anxiety, and post-traumatic stress disorder --all of which are risk factors for smoking. Smoking prevalence among women who have experienced IPV is as high as 51% to 70%. American Indian women, including Northern Plains Tribal women, experience the highest proportion of IPV among women from any racial/ethnic group. Furthermore, smoking prevalence among Northern Plains Tribal women is among the highest in the U.S. Specifically, among Northern Plains Tribal women who experienced IPV, 58% are current smokers. Multiple health interventions have been developed for women who have experienced IPV, including for alcohol and drug use given the high rates of these co-occurring problems. However, there have been no smoking cessation interventions among them. Trauma-informed, mindfulness-based approaches are shown to create physical, psychological, and emotional safety while mitigating habitual patterns of reactive or addictive behaviors by increasing awareness of reactivity and automated (e.g., smoking) behavior, allowing greater flexibility in response to cravings. These strength-based approaches are consistent with the values of American Indian culture and create opportunities for individuals who have been traumatized to rebuild a sense of choice and control. Our research team used an interactive, highly participatory approach to collect and use qualitative data to inform the initial development of a culturally tailored, trauma-informed smoking cessation intervention for Northern Plains Tribal women who have experienced IPV. Therefore, the primary objective of this application is to finalize the 8-session novel intervention and test its feasibility, acceptability, and satisfaction among a group of 48 Northern Plains Tribal women smokers who have experienced IPV. To achieve this goal, the following Aims will be addressed: 1) Use a community-based participatory approach with a Community Advisory Board to refine intervention materials and finalize the pilot intervention methodology; 2) Conduct a single arm intervention trial enrolling 48 Northern Plains Tribal women smokers who have experienced IPV to examine the primary study outcomes of feasibility, acceptability, and satisfaction with this culturally tailored, trauma-informed mindfulness smoking cessation intervention and the secondary study outcome of quit attempts and biochemically verified smoking abstinence prevalence at 3 and 6-months follow-up, which will gauge the effectiveness of the intervention; and 3) As an exploratory aim, the investigators will explore concurrent changes in drug and alcohol use given the proposed intervention's central focus on personal and historical trauma among American Indian women as contributors to addiction and consistent with a focus on poly- vs. single substance.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Report smoking ≥ 5 cigarettes per day
* A victim of physical and/or psychological IPV

Exclusion Criteria:

* Unable to provide informed consent
* < 18 years of age
* Plans on moving out of the region in the next six months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 3 years
  How feasible are our methods
Acceptability | 3 years
  How acceptable are our Methods to our participants
Satisfaction | 3 years
  How satisfactory are our methods with our participants

SECONDARY OUTCOMES:
Quit attempts | 3 years
  How many quit attempts did our participants make
Biochemically-verified smoking abstinence | 3 years
  Provide an estimate of this intervention's effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Nez Henderson, MD, MPH, Principal Investigator — Black Hills Center for American Indian Health
Locations (1):
- Black Hills Center for American Indian Health, Rapid City, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No